CLINICAL TRIAL: NCT07255560
Title: Clinical Evaluation of the Cosmetic Efficacy of the Product DMAE Oleate Aimed at Increasing Skin Firmness and Reducing Fine Lines and Wrinkles in Human Volunteers.
Brief Title: DMAE Oleate for Facial Skin Firmness and Fine Lines in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionos Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DMAE_Oleate_2025
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Skin Aging of Face and Hands; Facial Wrinkles - Rough Texture - Hyperpigmentation; Skin Laxity
Keywords: DMAE Oleate; Skin firmness; Fine lines & wrinkles; VISIA-CR imaging; Cutometer elasticity/fatigue
MeSH Terms: conditions — Cutis Laxa; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DMAE Oleate (Experimental): This group will be provided with the product DMAE Oleate.
  Interventions: Other: Topical DMAE Oleate

INTERVENTIONS:
Other: Topical DMAE Oleate — Volunteers will be provided with the product DMAE Oleate and instructed to apply one pump topically at night for 12 weeks (week 1: Monday, Wednesday, Friday, Sunday; weeks 2 to 12: nightly). Efficacy will be evaluated at baseline (D0) and at 4, 8, and 12 weeks using VISIA-CR® (crow's-feet wrinkle area/depth/volume), Cutometer® (firmness, elasticity, fatigue), and a self-assessment questionnaire. Product is supplied in individual containers and stored in a cool, dry place; a patch test has been performed for safety. All procedures occur at Bionos Biotech S.L. facilities.

SUMMARY:
This single-arm, cosmetic study will evaluate the efficacy of topical DMAE Oleate on facial skin firmness and lines/wrinkles in healthy adults. Thirty volunteers (40-55 years) will apply DMAE Oleate at night for 12 weeks (week 1: Monday/Wednesday/Friday/Sunday; weeks 2 to 12: nightly, one pump dose). Efficacy will be assessed at baseline, week 4, week 8, and week 12. The primary goals are to determine changes in fine lines/wrinkles at the crow's-feet region and biomechanical properties of the face skin. Wrinkle area, depth, and volume will be quantified by standardized VISIA-CR® image analysis, while firmness, elasticity, and fatigue will be measured with a Cutometer®. Participants will also complete a self-assessment questionnaire at each time point. Measurements are performed under identical conditions at all visits to enable within-subject comparisons from baseline.

DETAILED DESCRIPTION:
Skin aging reflects intrinsic and extrinsic processes that reduce collagen/elastin, diminish hyaluronic acid, and compromise firmness and elasticity, leading to fine lines and wrinkles. In this cosmetic study, investigators will assess the efficacy of topical DMAE Oleate on facial skin by quantifying changes in fine lines/wrinkles and biomechanical parameters of firmness, elasticity, and fatigue in healthy adult volunteers.

Thirty healthy volunteers aged 40-55 years with visible fine lines/wrinkles and signs of laxity/sagging will be enrolled at Bionos Biotech S.L. (Valencia, Spain) following informed consent and eligibility confirmation. Participants will receive DMAE Oleate in individual containers and will apply one pump topically once daily at night according to a fixed regimen: Week 1 on Monday, Wednesday, Friday, and Sunday; Weeks 2-12 nightly. Product handling and use will follow written instructions (apply to clean, dry facial skin; avoid the eye area; allow normal absorption before any other routine), and containers will be collected/verified at visits to support compliance documentation. All procedures and data processing will take place at Bionos Biotech facilities under standardized site conditions.

Assessments will be performed at baseline (D0), week 4 (D28), week 8 (D56), and week 12 (D84), in the same order at each visit to enable within-subject comparisons: (1) VISIA-CR® imaging of the crow's-feet region to quantify wrinkle area, depth, and volume; (2) Cutometer® measurements on facial skin to determine firmness, elasticity, and fatigue; and (3) completion of a self-assessment questionnaire. Participants will be reminded to maintain normal diet and hygiene, to refrain from initiating new/interfering cosmetics or oral supplements, to avoid excessive sun exposure and self-tanning/tanning salons, and to forgo intense or invasive cosmetic procedures for the study duration. The investigational product has undergone the required safety patch test prior to volunteer use; adverse events will be collected at each visit and managed according to site procedures. Volunteers must maintain normal diet and hygiene, refrain from starting new/interfering cosmetics or oral supplements, avoid excessive sun exposure and self-tanning/tanning salons, and forgo intense/invasive cosmetic treatments; contraception methods should remain unchanged from 6 weeks prior through study end. Key exclusions include sensitive skin; eczema/rosacea; pregnancy, breastfeeding, or planned pregnancy; and known allergy/sensitivity to product components.

The primary analysis will compare within-subject changes from baseline to post-treatment time points using paired t-tests or Wilcoxon signed-rank tests (two-sided α=0.05). A sample of 30 participants is expected, based on prior center experience, to detect ≈5-10% differences with 80% power, acknowledging that this is the first evaluation of this product.

Ethical conduct follows the Declaration of Helsinki, ICH guidelines, and local committee approvals; informed consent was obtained before any procedure. Data are coded and handled under Spanish data-protection law.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with visible signs of fine lines and wrinkles.
* Volunteers with visible signs of skin laxity/sagging.
* Informed of the purpose and the protocol of the study and signed a written informed-consent form.
* Additional criteria to be included by the client.

Exclusion Criteria:

* Volunteers with sensitive skin.
* Pre-existing skin conditions: Eczema, Rosacea.
* Pregnancy/breastfeeding/planning pregnancy.
* Known allergy/sensitivity to any component of the product.
* Agree to avoid excessive sun exposure/self-tanning product/avoid tanning salons/solariums.
* No lasers/tretinoin/procedures/facial hair removal/facials 2 weeks prior or during the study.
* Additional criteria to be included by the client.
* Any condition judged by the investigator to be unsuitable for participation in the study.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Quantification of the change in facial fine lines and wrinkles (crow's-feet) - area, depth, and volume - from baseline to post-treatment visits using VISIA-CR®. | Baseline (before product application) and after 4, 8, and 12 weeks of application.
  Thirty healthy volunteers (40-55 years) will apply topical DMAE Oleate for 12 weeks (week 1: Monday/Wednesday/Friday/Sunday at night; weeks 2 to 12: nightly, one pump). Standardized image capture with VISIA-CR® will be performed on the crow's-feet region at baseline (D0) and at 4 (D28), 8 (D56), and 12 weeks (D84) after application to compute wrinkle area, depth, and volume. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; product is supplied in individual containers, one-pump dose, stored cool and dry. A safety patch test has been completed prior to volunteer use.
Quantification of the skin firmness, elasticity, and fatigue from baseline to post-treatment visits using Cutometer®. | Baseline (before product application) and after 4, 8, and 12 weeks of application.
  Thirty healthy volunteers (40-55 years) will apply topical DMAE Oleate for 12 weeks (week 1: Monday/Wednesday/Friday/Sunday at night; weeks 2 to 12: nightly, one pump). Cutometer® measurements will be performed on facial skin to determine firmness, elasticity, and fatigue at baseline (D0) and at 4 (D28), 8 (D56), and 12 weeks (D84) after application. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; product is supplied in individual containers, one-pump dose, stored cool and dry. A safety patch test has been completed prior to volunteer use.
Completion of a self-assessment questionnaire. | Baseline (before product application) and after 4, 8, and 12 weeks of application.
  Thirty healthy volunteers (40-55 years) will apply topical DMAE Oleate for 12 weeks (week 1: Monday/Wednesday/Friday/Sunday at night; weeks 2 to 12: nightly, one pump). Participants will complete a self-assessment questionnaire at baseline (D0) and at 4 (D28), 8 (D56), and 12 weeks (D84) after application to provide a subjective evaluation of the treatment. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; product is supplied in individual containers, one-pump dose, stored cool and dry. A safety patch test has been completed prior to volunteer use.

CONTACTS AND LOCATIONS:
Overall Officials: Adela Serrano Gimeno, PhD, Principal Investigator — Bionos Biotech S.L. , LabAnalysis Life Science
Locations (1):
- Bionos Biotech S.L., LabAnalysis Life Science, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No